CLINICAL TRIAL: NCT06007482
Title: An Open-Label, Multicenter, First-in-Human, Phase 1 Study of ES009 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ES009 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elpiscience Biopharma Australia Pty. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Elpiscience Biopharma, Ltd. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES009-1001
Record Dates: First submitted 2023-08-10; First posted 2023-08-23 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor
Keywords: Leukocyte immunoglobulin-like receptor B2 (LILRB2)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation Cohort (Experimental): ES009 monotherapy dose level will be escalated in participants with advanced solid tumors.
  Interventions: Drug: ES009

INTERVENTIONS:
Drug: ES009 — ES009 is administered via intravenous infusion, once every 21 days.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of ES009 administered intravenously to subjects with advanced solid tumors.

DETAILED DESCRIPTION:
ES009 is a recombinant humanized IgG4 monoclonal antibody that specifically targets and blocks LILRB2. By reprograming suppressive myeloid cells into pro-inflammatory phenotypes, ES009 reshapes the immunosuppressive tumor microenvironment into an immune-favorable one to combat cancer development and progression.

This is a first-in-human, open-label, multicenter, non-randomized study designed to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD), optimal biological dose (OBD), and recommended phase 2 dose (RP2D) of ES009 by evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of ES009 administered intravenously to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Histological or cytological documentation of unresectable locally advanced or metastatic solid tumors, if 1) disease has progressed despite standard therapy, and no further standard therapy exists; or 2) standard therapy has proven to be ineffective or intolerable or is considered inappropriate.
* At least one measurable lesion per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* Life expectancy of at least 12 weeks.
* Adequate hematologic, hepatic, renal and coagulation function per protocol.
* Male and female subjects of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception per protocol.

Exclusion Criteria:

* Any prior therapy targeting LILRB2.
* Receipt of any investigational therapies within 28 days or 5 half-lives prior to the first dose of study drug.
* Prior treatment with the following therapies:• Anticancer therapy within 28 days or 5 half-lives of the drug prior to the first dose of study drug, whichever is shorter. Exception: hormonal replacement therapy.• A wash out of at least 2 weeks before the start of study drug for radiation to the extremities and 4 weeks for radiation to the chest, brain, or visceral organs is required.
* Prior allogeneic or autologous bone marrow transplantation or solid organ transplantation.
* Toxicity from previous anticancer treatment per protocol.
* Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug with certain exceptions.
* Subjects who received transfusion of blood products (including platelets or red blood cells), G-CSF, GM-CSF, recombinant erythropoietin, or recombinant thrombopoietin within 14 days prior to the first dose of study treatment.
* Major surgery within 4 weeks prior to the first dose of study treatment.
* Live vaccine therapies within 4 weeks prior to the first dose of study treatment.
* Recent history of allergen desensitization therapy within 4 weeks prior to the first dose of study treatment.
* Known allergies to CHO-produced antibodies.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last two years with certain exceptions.
* CNS metastases with certain exceptions.
* Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications.
* Active interstitial lung disease (ILD) or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
* Active infection requiring systemic therapy, known human immunodeficiency virus (HIV) infection, or positive test for hepatitis B active infection (HBsAg) or hepatitis C active infection (hepatitis C antibody).
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
* History or evidence of cardiac abnormalities.
* Pregnant or nursing females.
* Any known, documented, or suspected history of illicit substance abuse that would preclude subject from participation, unless clinically justified.
* Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illness/condition, which in the judgment of the Investigator might compromise the safety of the subject or integrity of the study, interfere with the subject participation in the trial or compromise the trial objectives.
* Involvement in the planning and/or conduct of the study (applies to both Sponsor/CRO staff and staff at the study site)
* Judgment by the Investigator that the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of adverse events of ES009 | 1-3 years
  Adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Maximum tolerated dose (MTD) of ES009 | 1-3 years
  The MTD of ES009 will be determined.
Optimal biological dose (OBD) of ES009 | 1-3 years
  The OBD of ES009 will be determined.
Recommended phase 2 dose (RP2D) of ES009 | 1-3 years
  The RP2D of ES009 will be determined.
Maximum administered dose (MAD) of ES009 | 1-3 years
  The MAD of ES009 will be determined.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of ES009 | 1-3 years
  Maximum observed serum concentration (Cmax) of ES009 will be measured.
Trough observed serum concentration (Ctrough) of ES009 | 1-3 years
  Trough observed serum concentration (Ctrough)of ES009 will be measured.
Area under the serum concentration time curve (AUC) of ES009 | 1-3 years
  Area under the serum concentration time curve (AUC) of ES009 will be measured.
Time to Cmax (Tmax) of ES009 | 1-3 years
  Time to Cmax (Tmax) of ES009 will be measured.
The terminal elimination half life of ES009 | 1-3 years
  The terminal elimination half-life (t 1/2) of ES009 will be measured.
Immunogenicity of ES009 | 1-3 years
  Frequency of anti-drug antibodies (ADA) against ES009 will be determined.
Preliminary antitumor activity of ES009 | 1-3 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Peninsula and South Eastern Oncology and Haematology Group, Frankston
  - St George Private Hospital, Kogarah
  - Scientia Clinical Research, Randwick
  - Sunshine Coast University Private Hospital, Sunshine Coast